CLINICAL TRIAL: NCT02949583
Title: Clinical Effectiveness and Microbiological Evaluation of a Mouthwash of Pomegranate (Punica Granatum Linn.) in School Children
Brief Title: Mouthwash of Pomegranate Against Biofilm and Gingival Inflammation in School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual da Paraiba (Other)
Responsible Party: Principal Investigator, DANÚBIA ROBERTA DE MEDEIROS NÓBREGA, Professor clinical, Universidade Estadual da Paraiba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Effectiveness of Pomegranate
Record Dates: First submitted 2014-05-20; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Gingivitis
Keywords: DENTAL PLAQUE; MEDICINAL PLANTS; GINGIVITIS
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Punica granatum Linn. (Experimental): The childrens used the mouthwash contain pomegranate 6,25% twice daily for 14 days.
  Interventions: Drug: Punica granatum Linn.
- chlorhexidine (Active Comparator): The childrens used the mouthwash contain chlorhexidine 0.12% twice daily for 14 days.
  Interventions: Drug: chlorhexidine

INTERVENTIONS:
Drug: Punica granatum Linn. — Mouthwash (6,25% of Punica granatum Linn) 10mL per day during 14 days
  Other Names: Pomegranate
  Arms: Punica granatum Linn.
Drug: chlorhexidine — standard anti-bacterial mouthwash Mouthwash (0,12% chlorhexidine) 10mL per day during 14 days
  Other Names: Periogard
  Arms: chlorhexidine

SUMMARY:
The mechanical control of supragingival biofilm is accepted as one of the most important measures to prevent dental caries and periodontal diseases. Nevertheless, maintaining dental surfaces biofilm-free is not an easy task. In this regard, numerous studies researches have demonstrated the effectiveness of mouthwashes containing antimicrobial active ingredients that prevent and control both supragingival biofilm and gingivitis, specially when used adjunctively to mechanical oral hygiene regimens.

DETAILED DESCRIPTION:
In vitro and clinical researches using Punica granatum Linn shows antimicrobial and antiadherent activity against dental biofilm microorganisms. The purpose of this study was to evaluate the clinical effectiveness of a mouthwash of Punica granatum Linn. against biofilm and gingival inflammation in school children

ELIGIBILITY:
Inclusion Criteria:

* Age group: 09-12 years old
* Presence of at least 20 teeth
* Simplified Oral Hygiene Index (S-OHI)≥ 1,6

Exclusion Criteria:

* Use of orthodontic appliance
* Recent (in the past 2 months)use of antibiotics and mouthwashes

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Difference in the Gingival Index scores. | Baseline, Seventh Day and Fourteeth day (14 days)
  On day 0, we measured the Plaque Index (PI) (Silness; Löe, 1964) at baseline, on the seventh day and on the fourteenth day.
Difference in the Gingival Bleeding Index scores. | Baseline, Seventh Day andFourteeth day (14 days)
  On day 0, we measured the Bleeding on Probing Index (BPI) (Ainamo; Bay, 1975) at baseline, on the seventh day and on the fourteenth day.
Difference in the Microbiological analysis of saliva for oral streptococcus count evolution from the start till the end of the study. | Baseline and Fourteeth day (14 days)
  At baseline, we collected non-stimulated saliva samples into a sterile container for counting of oral streptococci in the laboratory. And on the fourteenth day, we carried out the second saliva collection and measured the clinical indices used.

CONTACTS AND LOCATIONS:
Overall Officials: DANÚBIA RM NÓBREGA, Mastering, Principal Investigator — Universidade Estadual da Paraiba
Locations (1):
- Universidade Estadual Da Paraiba, Campina Grande, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menezes SM, Cordeiro LN, Viana GS. Punica granatum (pomegranate) extract is active against dental plaque. J Herb Pharmacother. 2006;6(2):79-92. PMID 17182487
- [Background] Bhadbhade SJ, Acharya AB, Rodrigues SV, Thakur SL. The antiplaque efficacy of pomegranate mouthrinse. Quintessence Int. 2011 Jan;42(1):29-36. PMID 21206931
- [Background] DiSilvestro RA, DiSilvestro DJ, DiSilvestro DJ. Pomegranate extract mouth rinsing effects on saliva measures relevant to gingivitis risk. Phytother Res. 2009 Aug;23(8):1123-7. doi: 10.1002/ptr.2759. PMID 19170139
- [Background] Vasconcelos LC, Sampaio FC, Sampaio MC, Pereira Mdo S, Higino JS, Peixoto MH. Minimum inhibitory concentration of adherence of Punica granatum Linn (pomegranate) gel against S. mutans, S. mitis and C. albicans. Braz Dent J. 2006;17(3):223-7. doi: 10.1590/s0103-64402006000300009. PMID 17262129